CLINICAL TRIAL: NCT02245815
Title: The Use of Probiotics (L. Acidophilus Boucardii vs. Multi-species) in the Prevention of Necrotizing Enterocolitis and Their Effect on Secreting IgA in the Feces of Premature Newborns Under Less Than 1500 g
Brief Title: Prevention of Necrotizing Enterocolitis of Premature Newborns Under Less Than 1500 g Using Probiotics
Acronym: (PEPP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Guadalupe Gómez Rodríguez, neonatologist, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-2013-1002-7
Record Dates: First submitted 2014-09-02; First posted 2014-09-22 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Infectious Diseases
Keywords: Necrotizing enterocolitis; Probiotics; Secreting IgA; Preterm newborns
MeSH Terms: conditions — Communicable Diseases; Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- use probiotics boucardii (Experimental): was administered the probiotic 1x10⁹ colonies forming units per day for 3 weeks
  Interventions: Dietary Supplement: use probiotics boucardii
- use probiotics Multi-species (Experimental): was administered the probiotic 1x10⁹ colonies forming units per day for 3 weeks
  Interventions: Dietary Supplement: use probiotics Multi-species

INTERVENTIONS:
Dietary Supplement: use probiotics boucardii — group A was administered the lactobacillus acidophilus boucardii probiotic (1x10⁹ colonies forming units (UFC) per day for 3 weeks). The diagnosis of (NEC) was made using the Bell criteria by the attending physician. Gastric tolerance was measured, the number and the characteristics of the feces before and after the administration of the probiotic, and also the levels of (IgA s) was measured at the beginning and at the end of treatment.
  Arms: use probiotics boucardii
Dietary Supplement: use probiotics Multi-species — Group B was administered multi-species probiotic (1x10⁹colonies forming units (UFC) per day for 3 weeks). The diagnosis of (NEC) was made using the Bell criteria by the attending physician. Gastric tolerance was measured, the number and the characteristics of the feces before and after the administration of the probiotic, and also the levels of (IgA s) was measured at the beginning and at the end of treatment.
  Arms: use probiotics Multi-species

SUMMARY:
The purpose of this study is to evaluate the incidence of necrotizing enterocolitis and its effect over the secreting immunoglobulin A in the feces with the use of probiotics of the strain Lactobacillus acidophilus boucardii vs. Multispecies in premature newborns weighting less than 1500 g.

DETAILED DESCRIPTION:
Randomized controlled trial, in the Neonatal department of Highly Specialized Medical Unit (UMAE) of Hospital Pediatric - Gynecology No. 48 of Mexican Institute of Social Security (IMSS ) on Leon, Mexico, between 15th of December 2013 and 30th of October 2014, on premature newborns of less than 1500 g. They were two groups of patients:

Group A: was given Lacteol fort, which contains 1x10⁹(CFU) of Lactobacillus acidophilus strain boucardii every 24 hours during 3 weeks. Its presentation is a powder of 160 mg. It's manufactured by (Carnot ® laboratories), scientific products .

Group B: was given multispecies probiotic, which contains 1x10⁹ (CFU) of Lactobacillus acidophilus, rhamnosus, casei, plantarum, Bifidobacterium infantis, Streptococcus thermophilus , every 24 hours during 3 weeks. Its presentation is a powder with 1. (ITALMEX laboratories), scientific products .

All patients received trophic enteral stimulation for 5 days, then an increasing amount of 12-20 ml/kg of breast milk on a daily basis, according to the Clinical Practice Guidelines of feeding premature newborns of the investigators hospital.

The envelops containing the probiotic they were labeled with patient data and handled to the nurse in charge of the feeding so that it can be added preferably to the prescribed breast milk, and administered at12 o´clock every day with the feeding.

The diagnosis of Necrotizing Enterocolitis (NEC) was made by the attending physician using Bell criteria. Moreover the attending physician did the adjustments in the amount of breast milk consumed by the patient.

Gastric tolerance will be observed through: the presence of vomit, abdominal distention, presence of blood or bile juice on the gastric tube, and the pattern and characteristics of the feces using a daily record.Stool samples were taken between 9 am. and 21:00., before the first administration of probiotics and at the end of the third week of probiotic treatment. The samples were processed and frozen at -70'C. Quantifying secrete immunoglobulin A (IgA s) was made by immunodiagnostic assay K8870, Benshein, Germany ELISA.

was monitored the clinical evolution of Necrotizing Enterocolitis (NEC), medical or surgical treatment and the complications.

ELIGIBILITY:
Inclusion Criteria:

* All of the premature newborns of 34 weeks of gestational age, and with a weight between 700 to 1500 g. that are admitted in the Neonatal Intensive Care Unit or the Neonatology Department that have no contraindication for oral intake in the first 7 days of life. Must not have been diagnosed of sepsis of early onset, prenatal asphyxia, patent ductus arterious with hemodynamic repercussion, major congenital malformations. In all cases the parents or legal guardian must sign the informed consent.

Exclusion Criteria:

* All preterm newborns younger than 34 weeks of gestational age that develop any disease different of (NEC) that require to stop the enteral feeding for more than seven days or whose parents or legal guardians revoke the informed consent form.

Ages: 27 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Gómez Rodríguez, M.D., Principal Investigator — University of Guanjuato
Locations (1):
- University of Guanajuato School of Medicine, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gomez-Rodriguez G, Amador-Licona N, Daza-Benitez L, Barbosa-Sabanero G, Carballo-Magdaleno D, Aguilar-Padilla R, Gonzalez-Ramirez E. Single strain versus multispecies probiotic on necrotizing enterocolitis and faecal IgA levels in very low birth weight preterm neonates: A randomized clinical trial. Pediatr Neonatol. 2019 Oct;60(5):564-569. doi: 10.1016/j.pedneo.2019.02.005. Epub 2019 Mar 2. PMID 30898471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: clinic
Groups:
- Use Probiotics Boucardii: group A will be administered the lactobacillus boucardii probiotic (1x109 colonies forming units (UFC) per day for 3 weeks).
  use probiotics Boucardii: group A will be administered the lactobacillus boucardii probiotic (1x109 colonies forming units (UFC) per day for 3 weeks). The diagnosis of NEC will be made using the Bell criteria by the attending physician. Gastric tolerance will be measured, the number and the characteristics of the feces before and after the administration of the probiotic, and also the levels of (IgA s) will be measured at the beginning and at the end of treatment.
- Use Probiotics Multi-species: Group B will be administered multi-species probiotic (1x109 colonies forming units (UFC) per day for 3 weeks).
  use probiotics Multi-species: Group B will be administered multi-species probiotic (1x109 colonies forming units (UFC) per day for 3 weeks). The diagnosis of NEC will be made using the Bell criteria by the attending physician. Gastric tolerance will be measured, the number and the characteristics of the feces before and after the administration of the probiotic, and also the levels of (IgA s) will be measured at the beginning and at the end of treatment.
Period: Overall Study
Arm/Group | Use Probiotics Boucardii | Use Probiotics Multi-species
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Use Probiotics Boucardii | Use Probiotics Multi-species | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45 | 45 | 90
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks of gestation] | 30.3 (1.83) | 31.1 (2.3) | 30.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  Mexico | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With (NEC)
Description: (NEC) was evaluated according to Bell's criteria and only considered in case of stage II-III
Time Frame: 3 weeks
Measure: Number; unit: participants
Groups:
- Probiotics Lactobacillus Acidophilus Boucardii: group A will be administered the Lactobacillus acidophilus boucardii probiotic (1x109 colonies forming units (UFC) per day for 3 weeks).
- Use Probiotics Multi-species: Group B will be administered multi-species probiotic (1x109 colonies forming units (UFC) per day for 3 weeks).
Arm/Group | Probiotics Lactobacillus Acidophilus Boucardii | Use Probiotics Multi-species
Number analyzed (Participants) | 45 | 45
participants | 0 | 1

2. Post Hoc Outcome: Change in Fecal Secretory IgA Levels From Baseline to 3 Weeks of Probiotics Use.
Description: The change was calculated from two time points (at 3 weeks of treatment minus baseline).
Time Frame: 3 weeks
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg/10g
Groups:
- Probiotics Lactobacillus Acidophilus Boucardii: Group A will be administered the Lactobacillus acidophilus boucardii probiotic
- Use Probiotics Multi-species: Group B will be administered multi-species probiotics
Arm/Group | Probiotics Lactobacillus Acidophilus Boucardii | Use Probiotics Multi-species
Number analyzed (Participants) | 45 | 45
mg/10g | 0.3 [0.15 to 0.45] | 0.56 [0.24 to 0.89]

ADVERSE EVENTS:
Time Frame: 11 months
Groups:
- Use Probiotics Lactobacillus Acidophilus Boucardii: group A will be administered the lactobacillus acidophilus boucardii probiotic (1x109 colonies forming units (UFC) per day for 3 weeks).
  use probiotics Lactobacillus acidophilus boucardii: group A will be administered the Lactobacillus acidophilus boucardii probiotic (1x109 colonies forming units (UFC) per day for 3 weeks). The diagnosis of NEC will be made using the Bell criteria by the attending physician. Gastric tolerance will be measured, the number and the characteristics of the feces before and after the administration of the probiotic, and also the levels of (IgA s) will be measured at the beginning and at the end of treatment.
Arm/Group | Use Probiotics Lactobacillus Acidophilus Boucardii | Use Probiotics Multi-species
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

LIMITATIONS AND CAVEATS:
The quantification of the amount of breast milk administered was imprecise because in the Unit there is no Milk Bank, and the visits from the mothers are restricted, however we acknowledge the crucial role of breast milk in the prevention of (NEC).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes